CLINICAL TRIAL: NCT03479125
Title: Protocol IDN-6556-18 - A Post Treatment Follow-up Study for Liver Disease Subjects With or Without Liver Cirrhosis After Receiving Emricasan or Placebo
Brief Title: Post-Treatment Follow-up Study for Liver Disease Subjects With or Without Cirrhosis After Receiving Emricasan or Placebo
Status: Terminated | Type: Observational
Why Stopped: Sponsor has discontinued the development of emricasan
Sponsor: Conatus Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: IDN-6556-18
Record Dates: First submitted 2018-03-20; First posted 2018-03-27 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Liver Diseases; Liver Fibrosis; Liver Cirrhosis; NASH Fibrosis; Decompensated Non-Alcoholic Steatohepatitis Cirrhosis; Orthotopic Liver Transplantation
MeSH Terms: conditions — Liver Diseases; Liver Cirrhosis | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Historical emricasan or placebo subjects: Subjects with liver fibrosis or cirrhosis who have received at least one dose of emricasan or placebo in a prior IDN-6556 study including IDN-6556-07, IDN-6556-12, IDN-6556-14 or IDN-6556-17.
  Interventions: Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Ultrasound — Subjects will be observed to estimate the adjusted event rate for hepatocellular carcinoma with or without cirrhosis previously treated with emricasan or placebo.
  Other Names: MRI. CT scan.

SUMMARY:
A post-treatment follow-up observational study for liver disease subjects with or without liver cirrhosis after receiving emricasan or placebo.

Subjects must have been enrolled in a prior IDN-6556 study to be eligible.

DETAILED DESCRIPTION:
A multi-center, post-treatment follow-up observational study for liver disease subjects with or without liver cirrhosis after receiving emricasan or placebo.

This phase 2 observational study will enroll subjects from Study IDN-6556-07 (Post Orthotropic Liver Transplantation - NCT02138253), IDN-6556-12 (NASH Fibrosis - NCT02686762), IDN-6556-14 (NASH Cirrhosis and Severe Portal Hypertension - NCT02960204) or IDN-6556-17 (Decompensated NASH Cirrhosis - NCT03205345) who have received at least one dose of emricasan or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects previously treated with at least 1 dose of emricasan or placebo from clinical studies IDN-6556-07 (post orthotopic liver transplant due to HCV), IDN-6556-12 (NASH fibrosis), IDN-6556-14 (NASH cirrhosis), or IDN-6556-17 (NASH cirrhosis).
2. Subjects able to provide written informed consent and able to understand and willing to comply with the requirements of the study.

Exclusion Criteria:

1. Use of controlled substances (including inhaled or injected drugs) or non-prescribed use of prescription drugs within 1 year of screening to the point of interfering with the subject's ability to comply, in the investigator's judgement, with study procedures.
2. Treatment with an investigational drug following treatment with emricasan or placebo.
3. Previous transplant unless subject was enrolled from IDN-6556-07 (post orthotopic liver transplant due to HCV).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who previously received at least one dose of emricasan or placebo in clinical study IDN-6556-07 (post orthotopic liver transplant due to HCV), IDN-6556-12 (NASH fibrosis), IDN-6556-14 (NASH cirrhosis), and IDN-6556-17 (NASH cirrhosis).
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Adjusted event rate for hepatocellular carcinoma. | 3 years
  To estimate the adjusted event rate for hepatocellular carcinoma in subjects with or without cirrhosis previously treated with emricasan or placebo.

SECONDARY OUTCOMES:
Adjusted event rate for all malignancies. | 3 years
  To estimate the adjusted event rate for all malignancies in subjects with or without cirrhosis previously treated with emricasan or placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Mason Yamashita, MD, Study Director — Conatus Pharmaceuticals Inc.
Locations (3):
- United States (3):
  - Inland Empire Liver Foundation, Rialto, California
  - Options Health Research, LLC, Tulsa, Oklahoma
  - Gastro One, Germantown, Tennessee